CLINICAL TRIAL: NCT04769063
Title: An Analysis of Kinesio® Tape on Mitigation of Dynamic Knee Valgus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Dakota State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB0003317
Record Dates: First submitted 2021-02-08; First posted 2021-02-24 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Knee Valgus
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hip (Experimental)
  Interventions: Other: Kinesio Tape
- Knee (Experimental)
  Interventions: Other: Kinesio Tape
- Control (No Intervention)

INTERVENTIONS:
Other: Kinesio Tape — Gluteus medius facilitation and knee spiral taping techniques will be applied to treat dynamic knee valgus
  Arms: Hip; Knee

SUMMARY:
Participants will completed a 5 minute warm-up on a stationary bike. Next, participants will perform 3 practice trials of the double leg jump landing (DJL) test off of a 30 cm box. In order for the trial to count the participants need to maintain their landing posture for at least 2 seconds, if they are unable to do so the trial will be repeated.

After the completion of three practice trials of the DJL test, the first taping condition will be applied. Each participant will receive 3 taping conditions to the dominant leg, a gluteus medius facilitation (GM), a spiral technique (ST), and no tape (NT). The order of conditions will be randomized.

The use of a no tape condition will act a control for both the jumping protocol and the Y-balance test. For this condition, no tape or intervention of any kind will be applied to the subject before completing either tasks. Regardless of the order of randomly assigned taping condition, the participant will rest 10 minutes in a non-weight bearing position before completing a round of testing.

During the 10-minute rest, 3D motion analysis sensors will be placed on the participant to assess hip internal rotation and knee valgus in the frontal plane. After the sensors are applied, the first follow-up Y Balance Test will be completed.

Each participant will complete the Y Balance Test 3 times, once for each condition. For the trial to count, the reach foot is not permitted to touch the floor and the hands have to remain stationary on the pelvis. If the participant fails to meet the testing criteria, the trial will be repeated. At the end of the trial, each testing direction distance will be written down and a mean score will be calculated.

Following the first Y balance test, three DJL tests will be performed, each separated by a 60-second rest period. Once the participant completes 3 approved trials, the first taping condition will be removed and the procedure will be repeated for the second and third taping procedures.

DETAILED DESCRIPTION:
The facilitative gluteus medius application was applied from origin to insertion of the muscle, as specified by Dr. Kase (2013). The subject was positioned in side-lying with the dominant leg facing up. The CKTP cut a Y-strip of Kinesio® Tex Classic Tape the same distance from the participant's ASIS to the greater trochanter of the femur. The tape was anchored at the ASIS with no tension followed by the participant moving into approximately 90° hip flexion, adduction, and internal rotation. Then, each tail of the Y-strip was applied at 25% tension towards the greater trochanter where it was anchored again with no tension. Following application, the participant was instructed to remain in a position of comfort for 10 minutes before continuing with the study protocol.

The second taping condition utilized is a spiral technique (ST), applied with Kinesio® Tex Performance Plus Tape. Participant positioning included standing in an open-packed, double-leg stance with feet approximately hip width apart. The CKTP anchored an I-strip of tape with no tension on the participant's medial aspect of the middle, tibia. With a stabilizing hand on the anchor, the practitioner pulled the tape with 75-100% tension and applied towards the lateral aspect of the tibiofemoral joint, Once the tape moved to the posterior side of the knee, the CKTP reduced the tension to 0% over the popliteal fossa so as to reduce skin tearing and provide another mechanism for pulling the knee out of valgum. When the tape crossed diagonally over the popliteal fossa, the CKTP again employed at 75-100% tension from the medial femoral condyle to the vastus lateralis. The tape was then secured to the posterior thigh with an anchor at 0% tension. Thus, the tape created a spiral shape up the participants' leg. Again, the subject was directed to rest comfortably in a non-weight bearing position for 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* current participation in basketball or volleyball

Exclusion Criteria:

* present pain with jumping or landing
* history of lower limb surgery within the12 months of the study
* any contraindications to Kinesio® Tape

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Three dimensional motion analysis | 1 day
  Assessment of knee valgus in the frontal plane
Y-balance test | 1 day
  Functional screening tool, which can be used to assess lower extremity stability, monitor rehabilitation progress, to understand deficits after injury, and identify athletes at high risk for lower extremity injury
Drop jump landing test | 1 day
  Clinical test with a high reliability of 95% to screen for lower limb injury, including a high specificity (46.07%) and sensitivity (95.04%) to predict ACL injury

CONTACTS AND LOCATIONS:
Locations (1):
- North Dakota State University, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No